CLINICAL TRIAL: NCT05921955
Title: Effect of Maternal Oxygen Supplementation by High-flow Nasal Oxygen Compared With Room Air on Fetal Acidemia
Brief Title: Application of High-flow Nasal Oxygen in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TREC2023-KY021
Record Dates: First submitted 2023-06-15; First posted 2023-06-27 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2023-04

CONDITIONS: Fetal Acidemia
Keywords: high-flow nasal oxygen; cesarean section; oxygen; umbilical artery; acidemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- air group (No Intervention): the patients of the air group receive the 2L/min with air pattern by the Optiflow high-flow nasal cannula system from anesthesia to fetal delivery.
- HFNO group (Experimental): For HFNO group, a flow rate of 40L/min, with 100% oxygen concentration and a temperature of 37℃ by the Optiflow high-flow nasal cannula system from anesthesia to fetal delivery.
  Interventions: Device: Optiflow high-flow nasal cannula system

INTERVENTIONS:
Device: Optiflow high-flow nasal cannula system — Using the Optiflow high-flow nasal cannula system to supply oxygen for maternal.
  Arms: HFNO group

SUMMARY:
The study propose that the using the high-flow nasl oxygen to provide oxygen for maternal can improve the fetal acidemia and the neonatal outcomes during cesarean section with combined spinal-epidural anesthesia.

DETAILED DESCRIPTION:
Maternal oxygen supplementation is widely used intrauterine resuscitation technique in clinical, which can improve fetal oxygenation and prevent fetal acidemia. The incidence of hypotension is high in cesarean section with combined spinal-epidural anesthesia. Hypotension contributes to insufficient perfusion of uterus and placenta, resulting in decreased fetal oxygen supply and neonatal acidemia. High flow nasal oxygen have a better improvement oxygenation of patients by providing high flow oxygen airflow with heating and humidification through nasal cannula.

ELIGIBILITY:
Inclusion Criteria:

* An elective cesarean section in Beijing Tongren Hospital
* ≥37 weeks' gestation
* American society of Aneshesiologists（ASA） I-III
* Aged 18 to 45 years old
* The fasting time is 6-8h, and the water restriction time is ≥2h
* Anesthesia: combined spinal-epidural anesthesia
* Agree to the study and sign the informed consent

Exclusion Criteria:

* Fetal or placental abnormalities are known
* Maternal has complications
* Maternal BMI ≥40 kg/m2
* History of difficult intubation or known difficult airway
* Contraindications for HFNO such as nasal lesions or structural changes
* Gastric reflux disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
umbilical artery lactate, mmol/L | the fetal delivery
  mmol/L

SECONDARY OUTCOMES:
umbilical artery pH value | the fetal delivery
  unitless
umbilical artery oxygen partial pressure(PO2) | the fetal delivery
  mmHg
umbilical artery partial pressure of carbon dioxide(PCO2) | the fetal delivery
  mmHg
umbilical artery base excess(BE), mmol/L | the fetal delivery
  mmol/L
the incidence of pH<7.20 and pH<7.10 | the fetal delivery
  percentage

CONTACTS AND LOCATIONS:
Overall Officials: guyan Wang, Study Director — Beijing Tongren Hospital
Locations (1):
- Beijing tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Raghuraman N, Temming LA, Doering MM, Stoll CR, Palanisamy A, Stout MJ, Colditz GA, Cahill AG, Tuuli MG. Maternal Oxygen Supplementation Compared With Room Air for Intrauterine Resuscitation: A Systematic Review and Meta-analysis. JAMA Pediatr. 2021 Apr 1;175(4):368-376. doi: 10.1001/jamapediatrics.2020.5351. PMID 33394020
- [Background] Qian G, Xu X, Chen L, Xia S, Wang A, Chuai Y, Jiang W. The effect of maternal low flow oxygen administration during the second stage of labour on umbilical cord artery pH: a randomised controlled trial. BJOG. 2017 Mar;124(4):678-685. doi: 10.1111/1471-0528.14418. PMID 28224745
- [Background] Raghuraman N, Wan L, Temming LA, Woolfolk C, Macones GA, Tuuli MG, Cahill AG. Effect of Oxygen vs Room Air on Intrauterine Fetal Resuscitation: A Randomized Noninferiority Clinical Trial. JAMA Pediatr. 2018 Sep 1;172(9):818-823. doi: 10.1001/jamapediatrics.2018.1208. PMID 30039159
- [Background] Zhou S, Cao X, Zhou Y, Xu Z, Liu Z. Ultrasound Assessment of Gastric Volume in Parturients After High-Flow Nasal Oxygen Therapy. Anesth Analg. 2023 Jul 1;137(1):176-181. doi: 10.1213/ANE.0000000000006340. Epub 2023 Jan 11. PMID 36630297
- [Background] Zhou S, Zhou Y, Cao X, Ni X, Du W, Xu Z, Liu Z. The efficacy of high flow nasal oxygenation for maintaining maternal oxygenation during rapid sequence induction in pregnancy: A prospective randomised clinical trial. Eur J Anaesthesiol. 2021 Oct 1;38(10):1052-1058. doi: 10.1097/EJA.0000000000001395. PMID 33259452
- [Derived] Li YH, Lei GY, Guo J, Yi M, Fu YJ, Wang GY. Effect of maternal oxygen supplementation for parturient undergoing elective cesarean section by high-flow nasal oxygen compared with room air on fetal acidemia: study protocol for a randomized controlled trial. Trials. 2024 Jan 22;25(1):73. doi: 10.1186/s13063-024-07927-y. PMID 38254137